CLINICAL TRIAL: NCT00668746
Title: Long-term Safety Evaluation of Minocycline Resistance After Treatment With Minocycline HCl Microspheres, 1 mg in Subjects With Chronic Periodontitis
Brief Title: Long-term Safety of Minocycline in Patients With Gum Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OraPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP-P-5756-1
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Periodontitis
Keywords: chronic periodontitis, antibiotic resistance
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline HCl microspheres (Experimental): Minocycline HCl microspheres
  Interventions: Drug: Minocycline HCl microspheres
- No drug intervention (No Intervention): No drug intervention

INTERVENTIONS:
Drug: Minocycline HCl microspheres — At Baseline and all interim visits, a single unit dose of 1mg minocycline HCl (with approximately 3mg PGLA) will be professionally administered subgingivally into periodontal pockets at each site exhibiting a PD ≥ 5mm.
  Other Names: minocycline
  Arms: Minocycline HCl microspheres

SUMMARY:
This study will look at the safety of using the study medicine for a long time. It will see if the germs get used to the medicine, making it not work as well, if it's used by people with gum disease for a long time.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the changes in populations of minocycline-resistant bacteria after long-term use of minocycline HCl microspheres, 1 mg in subjects with moderate-to-severe chronic periodontitis. This will be assessed through monitoring the total number and proportion of minocycline-resistant bacteria and the identity of minocycline-resistant species within a panel of 40 representative periodontal species in saliva and subgingival plaque.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* over 25 years of age
* moderate-to-severe chronic periodontitis
* documented informed consent
* willing to comply with contraceptive requirements
* free from any significant oral soft tissue pathology

Exclusion Criteria:

* willing to adhere to prohibitions and restrictions of the study
* oral health inappropriate for study inclusion
* females self-reporting pregnancy or lactation, or having a positive urine pregnancy result
* reporting any of the following conditions:

  * allergy to a tetracycline-class drug
  * systemic medical conditions requiring antibiotic prophylaxis prior to invasive dental procedures
  * active systemic infectious disease such as hepatitis, human immunodeficiency virus (HIV) or tuberculosis
  * diagnosed with clinically significant or unstable organic disease, or compromised healing potential, heart murmurs, histories of rheumatic fever, valvular disease or prosthetic joint replacement
* participation in a dental clinical trial or use of an investigational drug within 30 days of enrollment
* employees of the Investigator or study center, with direct involvement in the proposed study or other studies, as well as family members of the employees or the Investigator
* anyone who the investigator determines should not be included in the study for any reason that could compromise safety or the analysis of study results

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — OraPharma
Locations (1):
- Forsyth Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline HCl Microspheres: A single unit dose of 1mg minocycline HCl (with approximately 3mg PGLA) professionally administered subgingivally into periodontal pockets at each site exhibiting a PD ≥ 5mm
- No Drug Intervention: A control consisting of no drug intervention
Period: Overall Study
Arm/Group | Minocycline HCl Microspheres | No Drug Intervention
Started | 23 | 12
Completed | 21 | 11
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline HCl Microspheres | No Drug Intervention | Total
Number analyzed (Participants) | 23 | 12 | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 57.65 (10.71) | 52.83 (9.90) | 56.00 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 23 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Minocycline-Resistant Bacteria Using Bacterial Culture
Description: Percentage Change from Baseline is calculated as post-baseline percent minus baseline percent.
Time Frame: from Baseline to Day 30 and Day 180
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Minocycline HCl Microspheres | No Drug Intervention
Number analyzed (Participants) | 23 | 12
Percentage Change
  Plaque Sample at Day 30 | 13.15 (19.77) | 0.81 (3.33)
  Saliva Sample at Day 30 | 37.65 (113.9) | -2.25 (6.18)
  Plaque Sample at Day 180 | 8.09 (19.77) | 1.58 (2.49)
  Saliva Sample at Day 180 | 12.06 (18.35) | -0.51 (10.70)

2. Secondary Outcome: Micocycline-Resistance From Plaque Samples
Description: Percentage of Subjects showing Micocycline-Resistance for each Species from Plaque Samples DNA Method: Plaque Sample Intent-to-Treat Subjects - we report average of percentage for 4 plaque samples
Time Frame: Baseline, Day 30 and Day 180
Population: ITT
Measure: Number; unit: Percentage of Subjects
Arm/Group | Minocycline Group at Baseline | Minocycline Group at 30 Days | Micocycline Group at 180 Days | Control Group at Baseline | Control Group at 30 Days | Control Group at 180 Days
Number analyzed (Participants) | 23 | 23 | 23 | 12 | 12 | 12
Percentage of Subjects
  A.naeslundii | 7.14 | 1.19 | 17.86 | 6.82 | 6.82 | 13.64
  S.constellatus | 65.48 | 67.86 | 73.81 | 79.55 | 70.45 | 81.82
  E.nodatum | 3.57 | 3.57 | 13.10 | 11.36 | 6.82 | 13.64
  P.gingivalis | 29.76 | 21.43 | 7.14 | 29.55 | 15.91 | 2.27
  A.actinomucetemcomitans | 7.14 | 16.67 | 19.05 | 22.73 | 25.00 | 11.36
  F.nucleatum vincentii | 7.14 | 11.90 | 9.52 | 9.09 | 9.09 | 9.09
  C.rectus | 9.52 | 13.10 | 11.90 | 22.73 | 13.64 | 11.36
  R.dentocariosa | 0.00 | 2.38 | 5.95 | 9.09 | 9.09 | 2.27
  E.saburreum | 16.67 | 16.67 | 65.48 | 25.00 | 18.18 | 65.91
  P.micra | 8.33 | 15.48 | 23.81 | 29.55 | 22.73 | 9.09
  V.parvula | 41.67 | 71.43 | 53.57 | 47.73 | 54.55 | 31.82
  A.oris | 19.05 | 13.10 | 7.14 | 25.00 | 20.45 | 2.27
  S.anginosus | 30.95 | 30.95 | 34.52 | 50.00 | 59.09 | 50.00
  S.anguinis | 76.19 | 85.71 | 88.10 | 75.00 | 77.27 | 90.91
  A.gerencseriae | 3.57 | 10.71 | 2.38 | 6.82 | 6.82 | 0.00
  S.oralis | 70.24 | 78.57 | 82.14 | 77.27 | 79.55 | 88.64
  C.ochraccea | 1.19 | 0.00 | 1.19 | 2.27 | 0.00 | 0.00
  A.israelli | 0.00 | 2.38 | 2.38 | 2.27 | 0.00 | 0.00
  S.intermedius | 48.81 | 65.48 | 76.19 | 63.64 | 63.64 | 81.82
  C.matruchotti | 2.38 | 3.57 | 8.33 | 4.55 | 6.82 | 0.00
  P.nigrescens | 5.95 | 8.33 | 3.57 | 11.36 | 2.27 | 9.09
  A.odontolyticus | 4.76 | 19.05 | 21.43 | 25.00 | 20.45 | 9.09
  F.nucleatum polymorphum | 11.90 | 25.00 | 16.67 | 13.64 | 15.91 | 13.64
  C.showae | 4.76 | 10.71 | 7.14 | 34.09 | 15.91 | 15.91
  F.periodonticum | 1.19 | 9.52 | 2.38 | 2.27 | 0.00 | 0.00
  N.mucosa | 35.71 | 27.38 | 58.33 | 36.36 | 36.36 | 61.36
  F.nucleatum | 1.19 | 3.57 | 0.00 | 0.00 | 0.00 | 0.00
  C.ginigivaluis | 15.48 | 17.86 | 7.14 | 20.45 | 15.91 | 2.27
  S.gordonii | 72.62 | 91.67 | 69.05 | 81.82 | 75.00 | 77.27
  T.forsythia | 1.19 | 2.38 | 0.00 | 0.00 | 0.00 | 2.27
  S.noxia | 51.19 | 65.48 | 55.95 | 65.91 | 54.55 | 50.00
  P.acnes | 1.19 | 8.33 | 10.71 | 9.09 | 11.36 | 11.36
  P.melaninogenica | 7.14 | 3.57 | 2.38 | 2.27 | 2.27 | 13.64
  S.mitis | 75.00 | 79.76 | 75.00 | 81.82 | 77.27 | 90.91
  E.corrodens | 53.57 | 57.14 | 42.86 | 65.91 | 52.27 | 25.00
  G.morbillorum | 22.62 | 22.62 | 78.57 | 36.36 | 22.73 | 88.64
  C.sputigena | 1.19 | 0.00 | 3.57 | 4.55 | 0.00 | 4.55
  L.bucallis | 34.52 | 21.43 | 28.57 | 29.55 | 20.45 | 15.91
  C.gracilis | 7.14 | 4.76 | 4.76 | 4.55 | 0.00 | 0.00
  P.intermedia | 29.76 | 19.05 | 36.90 | 27.27 | 18.18 | 31.82

3. Secondary Outcome: Micocycline-Resistance From Saliva Sample
Description: Percentage of Subjects Showing Micocycline-Resistance for each Species from Saliva Sample DNA Method: Saliva Sample Intent-to-treat Subjects
Time Frame: Baseline, Day 30 and Day 180
Population: ITT
Measure: Number; unit: Percentage of Subjects
Arm/Group | Minocycline Group at Baseline | Minocycline Group at Day 30 | Minocycline Group at Day 180 | Control Group at Baseline | Control Group at Day 30 | Control Group at Day 180
Number analyzed (Participants) | 23 | 23 | 23 | 12 | 12 | 12
Percentage of Subjects
  A.naeslundii | 4.76 | 0.00 | 19.05 | 9.09 | 9.09 | 0.00
  S.constellatus | 47.62 | 42.86 | 80.95 | 72.73 | 63.64 | 63.64
  E.nodatum | 4.76 | 0.00 | 14.29 | 9.09 | 0.00 | 9.09
  P.gingivalis | 23.81 | 19.05 | 9.52 | 27.27 | 18.18 | 18.18
  A.actinomucetemcomitans | 19.05 | 9.52 | 14.29 | 27.27 | 0.00 | 27.27
  F.nucleatum vincentii | 9.52 | 0.00 | 19.05 | 9.09 | 0.00 | 18.18
  C.rectus | 9.52 | 9.52 | 14.29 | 18.18 | 0.00 | 0.00
  R.dentocariosa | 4.76 | 0.00 | 14.29 | 9.09 | 0.00 | 9.09
  E.saburreum | 19.05 | 14.29 | 61.90 | 27.27 | 0.00 | 72.73
  P.micra | 14.29 | 9.52 | 23.81 | 18.18 | 0.00 | 18.18
  V.parvula | 61.90 | 90.48 | 80.95 | 81.82 | 81.82 | 90.91
  A.oris | 14.29 | 14.29 | 14.29 | 27.27 | 18.18 | 9.09
  S.anginosus | 14.29 | 14.29 | 42.86 | 27.27 | 9.09 | 45.45
  S.anguinis | 61.90 | 85.71 | 100.00 | 72.73 | 72.73 | 100.00
  A.gerencseriae | 4.76 | 14.29 | 9.52 | 9.09 | 0.00 | 9.09
  S.oralis | 66.67 | 71.43 | 100.00 | 63.64 | 90.91 | 90.91
  C.ochraccea | 0.00 | 0.00 | 4.76 | 9.09 | 0.00 | 0.00
  A.israelli | 0.00 | 0.00 | 0.00 | 9.09 | 0.00 | 0.00
  S.intermedius | 42.86 | 38.10 | 80.95 | 63.64 | 45.45 | 90.91
  C.matruchotti | 9.52 | 9.52 | 23.81 | 9.09 | 9.09 | 36.36
  P.nigrescens | 9.52 | 4.76 | 0.00 | 0.00 | 0.00 | 0.00
  A.odontolyticus | 23.81 | 19.05 | 28.57 | 45.45 | 0.00 | 36.36
  F.nucleatum polymorphum | 19.05 | 19.05 | 14.29 | 9.09 | 9.09 | 27.27
  C.showae | 19.05 | 9.52 | 4.76 | 36.36 | 0.00 | 9.09
  F.periodonticum | 4.76 | 4.76 | 4.76 | 9.09 | 0.00 | 0.00
  N.mucosa | 47.62 | 28.57 | 76.19 | 36.36 | 27.27 | 72.73
  F.nucleatum | 0.00 | 0.00 | 9.52 | 0.00 | 0.00 | 9.09
  C.ginigivaluis | 23.81 | 9.52 | 19.05 | 18.18 | 0.00 | 9.09
  S.gordonii | 71.43 | 85.71 | 66.67 | 72.73 | 45.45 | 72.73
  T.forsythia | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00
  S.noxia | 52.38 | 52.38 | 57.14 | 54.55 | 54.55 | 72.73
  P.acnes | 9.52 | 9.52 | 19.05 | 9.09 | 0.00 | 27.27
  P.melaninogenica | 0.00 | 0.00 | 19.05 | 18.18 | 18.18 | 0.00
  S.mitis | 61.90 | 71.43 | 90.48 | 81.82 | 90.91 | 100.00
  E.corrodens | 57.14 | 47.62 | 57.14 | 72.73 | 81.82 | 45.45
  G.morbillorum | 38.10 | 14.29 | 76.19 | 27.27 | 0.00 | 100.00
  C.sputigena | 9.52 | 4.76 | 0.00 | 9.09 | 0.00 | 0.00
  L.bucallis | 33.33 | 23.81 | 38.10 | 18.18 | 9.09 | 27.27
  C.gracilis | 0.00 | 0.00 | 4.76 | 0.00 | 0.00 | 0.00
  P.intermedia | 23.81 | 19.05 | 33.33 | 18.18 | 27.27 | 54.55

ADVERSE EVENTS:
Time Frame: 180 Days
Arm/Group | Minocycline HCl Microspheres | No Drug Intervention
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/12
Other Adverse Events (participants affected / at risk) | 8/23 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline HCl Microspheres (N=23) | No Drug Intervention (N=12)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline HCl Microspheres (N=23) | No Drug Intervention (N=12)
SINUSITIS (Infections and infestations) | 2 (2) | 0 (0)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 1 (1)
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 2 (2) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No